CLINICAL TRIAL: NCT04822675
Title: A Prospective Randomized Trial Comparing the Surgical Treatment of Ischemic Mitral Regurgitation Versus Percutaneous Mitral Repair Followed by Surgical Revascularization
Brief Title: REvascularization and Valve Intervention for Ischemic Valve diseasE: REVIVE Trial
Acronym: REVIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20210317
Record Dates: First submitted 2021-03-25; First posted 2021-03-30 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Mitral Valve Insufficiency; Coronary Artery Disease
MeSH Terms: conditions — Mitral Valve Insufficiency; Coronary Artery Disease | interventions — Replantation

STUDY DESIGN:
Intervention Model Description: Prospective randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous mitral repair (Experimental): Percutaneous mitral repair +/- coronary artery bypass grafting within 14 days of mitral repair.
  Interventions: Procedure: Percutaneous mitral valve repair
- Mitral valve surgery (Active Comparator): Surgical mitral valve surgery +/- coronary artery bypass grafting
  Interventions: Procedure: Surgical mitral valve repair/replacement

INTERVENTIONS:
Procedure: Percutaneous mitral valve repair — Percutaneous mitral repair will be performed using the MitraClip system.
  Arms: Percutaneous mitral repair
Procedure: Surgical mitral valve repair/replacement — All mitral valve surgeries will be performed either via sternotomy or right thoracotomy, and with cardioplegic arrest and cardiopulmonary bypass. Mitral valve repair may include annuloplasty and adjunctive procedures as determined by the operating surgeon. For mitral valve replacement, the choice of mitral valve prosthesis will be left at the surgeon's discretion.
  Arms: Mitral valve surgery

SUMMARY:
Ischemic mitral regurgitation (MR) and coronary artery disease is common and associated with significant morbidity and mortality. Ischemic MR has been traditionally treated surgically through either valve repair or replacement at the time of concomitant bypass grafting. Although patients with ischemic MR represent a heterogeneous group, outcomes for these patients over the intermediate term is poor owing to left ventricle (LV) dysfunction causing MR and the presence of coronary disease, which portends poor survival. There is an emergence of percutaneous therapies to treat MR which have been shown to be a less invasive, safe, and viable approach to treat comorbid patients.

The decision to treat ischemic MR either surgically or percutaneously is influenced by the presence of coronary disease and the ability to provide adequate revascularization. Mitral valve surgery concomitant to surgical revascularization, however, is associated with a several fold increase in mortality. In fact, the incremental risk increase is further magnified in high-risk patients. We therefore propose a novel prospective study to guide intervention for ischemic MR. Patients will be randomized to undergo surgical therapy with either mitral repair/replacement and/or concomitant coronary artery bypass grafting OR percutaneous mitral repair, followed by coronary artery bypass grafting.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with severe ischemic Mitral regurgitation (MR), as defined by the 2017 American Society of Echocardiography (ASE) guidelines for noninvasive evaluation of native valvular regurgitation.
2. Presence of reversible myocardial ischemia confirmed by preoperative myocardial viability study using radionuclide imaging.

Exclusion Criteria:

1. Patients with mixed mitral valve pathology, including fibroelastic deficiency, rheumatic valve disease, ruptured mitral valve chordae, mitral valve endocarditis.
2. Patients with acute ischemic MR, defined as MR caused by papillary muscle infarction and rupture.
3. Age < 18 years.
4. Prohibitive surgical risk or contraindications to Cardiopulmonary bypass (CPB) as defined by the Heart Team.
5. Need for a concomitant surgical procedure, excluding Coronary artery bypass grafting (CABG), tricuspid valve repair, Patent foramen ovale (PFO) closure, Atrial septal defect (ASD) closure and Maze procedure.
6. Prior mitral valve repair procedure (percutaneous or surgical).
7. Leaflet anatomy unsuitable for MitraClip implantation, proper MitraClip positioning on the leaflets or sufficient reduction in MR by the MitraClip.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-08-12 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Mortality rate | Within 12 months of intervention
  All-cause mortality. Death from cardiovascular and non-cardiovascular causes.
Rate of myocardial infarction | Within 12 months of intervention
  These will be defined according to the Fourth Universal Definition of Myocardial Infarction
Rate of Stroke | Within 12 months of intervention
  1) New, acute focal neurological deficit thought to be of vascular origin with signs or symptoms lasting > 24 h and confirmed by a neurologist or 2) new, focal neurological deficit lasting > 24 h with imaging evidence of cerebral infarction or intracerebral hemorrhage.
Hospitalization rate for congestive heart failure | Within 12 months of intervention
  Admission to hospital with congestive heart failure exacerbation being the primary reason for admission. Congestive heart failure exacerbation is defined as 1) evidence of fluid overload and elevated filling pressures (for example, a central venous pressure > 8mmHg and/or a pulmonary capillary wedge pressure > 18mmHg) and/or 2) new decrease in cardiac output (for example, cardiac index < 2.2 L/min/m2) and end-organ perfusion (measured by one or more of: urine output < 20mL/hr, lactate >= 2.0, mixed venous oxygen saturation < 70%).

SECONDARY OUTCOMES:
Change in indexed left atrial volume | Within 6 and12 months of intervention
Degree of left ventricular remodeling | Within 6 and12 months of intervention
  Quantified by the change in left ventricular end systolic volume index
Presence of recurrent MR ≥2+ | Within 6 and12 months of intervention
  Defined as a regurgitant volume of 30-44 ml, a right ventricular ejection fraction of 30-39%, or an effective regurgitant orifice area of 20-29 mm2
Rate of mitral valve re-intervention | Within12 months of intervention
Number of Participants with worsening in heart failure symptoms | Within 6 and12 months of intervention
  +1 NYHA Class
Cumulative hospital days | Within 12-months of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Chan, MD, MPH, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada